CLINICAL TRIAL: NCT04958707
Title: Evaluating the Feasibility of a Mobile Phone-based Intervention (Zalo App) on Depression, Anxiety, and Stress of Family Caregivers of People With Dementia.
Brief Title: A Mobile Phone-based Intervention on Dementia Patients' Caregivers in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Collaborators: National Geriatric Hospital (Other Government); University of California, Davis (Other)
Responsible Party: Principal Investigator, Nguyen Tran To Tran, Lecturer of Geriatrics Department, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AG064688
Record Dates: First submitted 2021-06-20; First posted 2021-07-12 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Phase 1: 20 in-depth interviews to determine what knowledge and skills related to dementia patient care the carers need providing Phase 2: 60 carers will be randomly allocated into the interventional or controlled group. The intervention duration will be 8 weeks with providing knowledge and skills related to patient care.
Who Masked: Investigator
Masking Description: The investigator who interview the participants will be blinded during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informational support group (Experimental): The participants in the intervention group will be added to a chat group in the Zalo app, created and managed by one investigator, which is named The Dementia Caregiver Support group. Weekly, the investigator will post one of the topics identified in Phase 1. Before posting the information, the investigator will ask the participants what topic they would like to read and discuss the week after by voting the answer. The posted information will be based on evidence-based resources and consulted by geriatricians, the neurologist, and the psychologist who specialize in dementia. Immediately after posting the topic, one investigator will call the participants to ensure they read and understand the post. The chat group monitor will also collect the questions or comments from the carers who are encouraged to share their feelings or experiences with relevant questions. Then the monitor will post the answers after consulting with the experts.
  Interventions: Other: Information including knowledge and skills related to dementia patient care
- Controlled group (Active Comparator): The participants will receive usual care, introduced to the website Alzheimer.org to search for eligible information.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Information including knowledge and skills related to dementia patient care — The intervention will be administered to the participants via a smartphone app (Zalo app). Weekly, the investigator will post one of the eight topics identified in Phase 1 in the chat room. After posting the topic, one investigator will call the participants to ensure they read and understand the contents.
  Arms: Informational support group
Other: Usual care — Caregivers will be introduce to the website www.alzheimer.org to search for eligible information
  Arms: Controlled group

SUMMARY:
Background: The growing number of older people with dementia increases demand on informal caregivers who lack information and skills, leading to a high psychological burden in care provision. The proposed smartphone app-based intervention will provide a convenient and feasible solution for reducing depression, stress, and anxiety among dementia carers in Vietnam. This study aims to: (1) understanding the information and skills required by informal carers to populate the content of the intervention and (2) test the clinical feasibility of the intervention and feasibility of a fully- power randomized controlled trial.

Methods: The setting of this study is the geriatrics department in Gia Dinh People's hospital in Ho Chi Minh City. The eligible participants are the informal caregivers of patients with dementia living in the community, who use smartphones. Phase 1 will involve 20 interviews, conducted with 20 dementia carers to determine what information and skills they need most. These findings will be used to design the content of the intervention, which will comprise 8 weekly, online, psycho-educational, group sessions hosted on the Zalo app. Phase 2: using a pilot randomized control trial design, 60 participants will be assigned to the intervention or control group by the block randomization method with a ratio of 1:1. The participants will complete questionnaires at baseline, post-intervention and 3 month post-intervention. Outcome measures include DASS21 (Depression, anxiety and stress 21), dementia understanding, perceived social support, and caregiver's perceived burden. The primary outcome is the feasibility of the intervention and a future fully-power randomized controlled trial including acceptability and perceived effectiveness of the intervention and the rate of recruitment, retention, and completion of assessments.

DETAILED DESCRIPTION:
The study has two phases: the co-design of the content of the intervention (phase 1) and the randomized controlled trial phase (phase 2). The setting and the participants' eligibility criteria are the same for the two phases.

Phase 1 Design: a qualitative study will be conducted on 20 caregivers of patients with dementia to identify what information they most require.

Method: 20 face-to-face interviews will be held and guided by a trained geriatrician, in a private room in the geriatrics department. The open-ended questions are used, including "what difficulties are the participant facing in taking care of the patient with dementia?", "what information do the participant need most?". Each participant will be free to share thoughts. The interviews will be audio-recorded and fully transcribed.

Data analysis: The investigator will use inductive thematic content analysis. The eight most common issues in which the carers need providing information will be determined to shape for the intervention in phase 2.

Phase 2 Study design A parallel-group randomized controlled pilot trial will be used with equal randomization of 1:1 to test the feasibility and the acceptability of the smartphone app-based intervention. Sixty dementia carers, who meet the eligible criteria and are provided written informed consent, will be enrolled in the study and will be allocated to the intervention or usual care group.

Randomization The eligible participants will be assigned to the intervention or control group by an independent statistician, using the block randomization method (blocks of 4).

Intervention The participants in the intervention group will be added to a chat room in the Zalo app, created and managed by one investigator, which is named The Dementia Caregiver Support group. Weekly, the investigator will post one of the eight topics identified in Phase 1. Before posting the information, the investigator will ask the participants what topic they would like to read and discuss the week after by voting the answer. The posted information will be based on evidence-based resources and consulted by geriatricians, the neurologist, and the psychologist who specialize in dementia. Immediately after posting the topic, one investigator will call the participants to ensure the participants read and understand the post. The chat group monitor will also collect the questions or comments from the carers who are encouraged to share feelings or experiences with relevant questions. Then the investigator will post the answers after consulting with the experts.

Usual care: The participants in the control group will be introduced to the website Alzheimer.org to search for eligible information Procedure The characteristics of the participants (age, gender, educational level, relationship to the care recipient, time of care, etc.) and other assessments will be collected by an independent investigator, who will be blinded through the study.

Measures The participants will perform the Depression, anxiety and stress scale 21 (DASS21) questionnaire via phone call interviews. DASS21 scale contains 21 items, evaluating 3 subscales including depression, anxiety, and stress states over the past week. Higher scores indicate more severity of emotional states. Dementia understanding of the participants will be evaluated at baseline and post-intervention by a questionnaire, originating from the Northern Ireland Life and Time Survey, which was translated into Vietnamese. This questionnaire contains 7 items, for example, "dementia is a normal part of aging" or "dementia can be cured". The response options will be completed with yes/no choices. Four or fewer correct answers will be coded as low understanding, five correct answers medium understanding, and six or more answers as high understanding.

Perceived social support will be assessed using the Multidimensional Scale of Perceived Social Support (MSPSS), comprising 12 self-report items assessing the perceived support from family, friends, or significant others (eg, "There is a person who is around me when I am in need). Each item is scored from 1 (very strongly disagree) to 7 (very strongly agree), based on a 7-point Likert scale. Higher scores indicate higher degrees of perceived social support. This scale will be translated and adapted into Vietnamese.

The caregiver's perceived burden will be evaluated usingthe Zarit 4-item burden interview. Each item is scored from 0 to 4, and higher scores indicate higher levels of burden.

Outcome measurements will be assessed face-to-face at baseline and via phone calls at immediate post-intervention and 3-month follow-up post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being the primary caregivers of patients with dementia for at least the past 6 months and will continue to be for the next 6 months of the intervention. Dementia patients are those who have been diagnosed with dementia for at least 6 months and are living in the community.
* Being able to read and understand Vietnamese (at least primary education), and willing to participate in the study.
* Having a smartphone that has the Zalo app or willing to have this Zalo app be installed (there will be short training of using Zalo for new users)
* Aged ≥ 18 years

Exclusion Criteria:

* Having any acute diseases or cognitive impairment (screening by Mini-Cog),
* Having vision or hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: The Than, Dr, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (2):
- Vietnam (2):
  - Gia Dinh People's Hospital, Ho Chi Minh City
  - University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No
Share the results of the study

REFERENCES:
- [Result] McParland P, Devine P, Innes A, Gayle V. Dementia knowledge and attitudes of the general public in Northern Ireland: an analysis of national survey data. Int Psychogeriatr. 2012 Oct;24(10):1600-13. doi: 10.1017/S1041610212000658. Epub 2012 May 17. PMID 22591515
- [Result] Bruwer B, Emsley R, Kidd M, Lochner C, Seedat S. Psychometric properties of the Multidimensional Scale of Perceived Social Support in youth. Compr Psychiatry. 2008 Mar-Apr;49(2):195-201. doi: 10.1016/j.comppsych.2007.09.002. Epub 2007 Dec 21. PMID 18243894
- [Result] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Result] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- See also: The questionnaire will be used to evaluate dementia understanding of caregivers — https://pubmed.ncbi.nlm.nih.gov/22591515/
- See also: The questionnaire will be used to evaluate perceived social support — http://pubmed.ncbi.nlm.nih.gov/18243894/
- See also: The questionnaire will be used to evaluate stress and coping style — https://pubmed.ncbi.nlm.nih.gov/9988301/
- See also: DASS21 questionnaire will be used in depression, anxiety and stress — https://pubmed.ncbi.nlm.nih.gov/7726811/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1 (Qualitative interviews): Twenty qualitative interviews were conducted to explore the needs of caregivers of people with dementia.
  Phase 2 (Pilot RCT): We invited 60 eligible participants, who were then randomly assigned to either the control or intervention group.
Groups:
- Phase 2: Informational Support Group (Intervention Group): The participants in the intervention group will be added to a chat group in the Zalo app, created and managed by one investigator, which is named The Dementia Caregiver Support group. Weekly, the investigator will post one of the topics identified in Phase 1. Before posting the information, the investigator will ask the participants what topic they would like to read and discuss the week after by voting the answer. The posted information will be based on evidence-based resources and consulted by geriatricians, the neurologist, and the psychologist who specialize in dementia. Immediately after posting the topic, one investigator will call the participants to ensure they read and understand the post. The chat group monitor will also collect the questions or comments from the carers who are encouraged to share their feelings or experiences with relevant questions. Then the monitor will post the answers after consulting with the experts.
- Phase 2: Control Group: The participants will receive usual care, introduced to the website Alzheimer.org to search for eligible information.
- Phase 1: Qualitative Interviews: Twenty qualitative interviews were conducted to explore the needs of caregivers of people with dementia.
Period: Post Intervention
Arm/Group | Phase 2: Informational Support Group (Intervention Group) | Phase 2: Control Group | Phase 1: Qualitative Interviews
Started | 30 | 30 | 20
Completed | 29 | 30 | 20
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: 3 Months Follow- up
Arm/Group | Phase 2: Informational Support Group (Intervention Group) | Phase 2: Control Group | Phase 1: Qualitative Interviews
Started | 29 | 30 | 0 (The participants in Phase 1 were not followed up further)
Completed | 27 | 27 | 0 (The participants in Phase 1 were not followed up further)
Not Completed | 2 | 3 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Qualitative Interviews: The needs for knowledge and caregiving skills in dementia care were explored through in-depth interviews
- Phase 2: Informational Support Group (Intervention Group): Participants in the intervention group will be added to a chat group on the Zalo smartphone app, named The Dementia Caregiver Support Group. This group will be created and managed by one of the investigators. Each week, the investigator will post one of the eight topics identified in Phase 1. Prior to each post, participants will be invited to vote on which topic they would like to read and discuss the following week.
  The educational content shared will be based on evidence-based resources and reviewed by specialists, including geriatricians, a neurologist, and a psychologist with expertise in dementia care. Immediately after posting, the investigator will contact each participant to ensure that they have read and understood the content.
  Participants will be encouraged to share their feelings, experiences, and questions in the chat group. The investigator will monitor the chat, collect comments and questions, and post expert-reviewed responses.
  The intervention will last for seven weeks, covering seven topics: Feeding and incontinence care; Managing behavioral changes; Pressure injury prevention and care; Fall prevention; Understanding dementia progression; Preparing caregivers for future care; Caregiver self-care
- Phase 2: Control Group: The participants will receive usual care and be introduced to the website Alzheimer.org to search for eligible information.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Qualitative Interviews | Phase 2: Informational Support Group (Intervention Group) | Phase 2: Control Group | Total
Number analyzed (Participants) | 20 | 30 | 30 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (10.1) | 56.1 (10.1) | 54.1 (8.1) | 55.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 24 | 65
  Male | 2 | 7 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 30 | 30 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 20 | 30 | 30 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Vietnam | 20 | 30 | 30 | 80
Marital status [Count of Participants; unit: Participants]
  Having a partner | 12 | 16 | 19 | 47
  Single/widowed/divorce | 8 | 14 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: The Most Common Topics Related to Dementia Patient Care Skills
Description: The investigators will address these issues by in-deep interviews in phase 1. The most common topics the participants need providing will be listed
Time Frame: 4 months
Measure: Number; unit: Participants
Groups:
- The Information Needed by the Caregivers: We conducted in-depth interviews with 20 caregivers to identify the information and skills they need while providing care.
Arm/Group | The Information Needed by the Caregivers
Number analyzed (Participants) | 20
Participants
  Providing personal care | 15
  Managing behavior changes in care recipients. | 12
  Help-seeking strategies for caregivers | 18
  Self-care for caregivers to maintain their own well-being | 18
  Dementia progress and caring skills | 17
  Managing comorbidities such as pressure injuries, falls, and infections in care recipients | 15

2. Primary Outcome: Phase 2: The Rate of Recruitment, Retention and Completeness of Outcome Measurements
Description: The rate of recruitment will be identified by the percentage of participants who agree to participate in the study.
  The rate of retention will be identified by the percentage of participants who stay in the study. The rate of completeness of the outcome measurements is the percentage of participants who agreed to answer the questionnaires during the study. The rate of recruitment, the rate of participant retention, and the rate of completeness of outcome measurements will be reported in percentages.
Time Frame: 9 months
Measure: Number; unit: participants
Groups:
- Informational Support Group: The participants in the intervention group will be added to a chat room in the Zalo app, created and managed by one investigator, which is named The Dementia Caregiver Support group. Weekly, the investigator will post one of the topics identified in Phase 1. Before posting the information, the investigator will ask the participants what topic they would like to read and discuss the week after by voting the answer. The posted information will be based on evidence-based resources and consulted by geriatricians, the neurologist, and the psychologist who specialize in dementia. Immediately after posting the topic, one investigator will call the participants to ensure the participants read and understand the post. The chat group monitor will also collect the questions or comments from the carers who are encouraged to share feelings or experiences with relevant questions. Then the investigator will post the answers after consulting with the experts.
- Control Group: The participants in the control group will be introduced to the website Alzheimer.org to search for eligible information
Arm/Group | Informational Support Group | Control Group
Number analyzed (Participants) | 31 | 31
participants
  The recruitment rate | 30 | 30
  Retention rate | 27 | 27
  Completeness of outcome measurements | 27 | 27

3. Secondary Outcome: Phase 2: Depression, Anxiety and Stress Levels of the Caregivers
Description: The participants will be evaluated by the Depression, anxiety, and stress 21 scale. The minimum score is 0, and the maximum score is 126. The higher scores indicate worse outcome
Time Frame: Baseline, post-intervention (6 months) and three-month follow-up (9 months)
Population: In the intervention group, one participant withdrew during the intervention, and two participants withdrew after the intervention.
  In the control group, three participants were lost to follow-up.
Measure: Mean (Standard Error); unit: points
Groups:
- Informational Support Group (Intervention Group): The participants in the intervention group will be added to a chat room in the Zalo app, created and managed by one investigator, which is named The Dementia Caregiver Support group. Weekly, the investigator will post one of the topics identified in Phase 1. Before posting the information, the investigator will ask the participants what topic they would like to read and discuss the week after by voting the answer. The posted information will be based on evidence-based resources and consulted by geriatricians, the neurologist, and the psychologist who specialize in dementia. Immediately after posting the topic, one investigator will call the participants to ensure the participants read and understand the post. The chat group monitor will also collect the questions or comments from the carers who are encouraged to share feelings or experiences with relevant questions. Then the investigator will post the answers after consulting with the experts.
Arm/Group | Informational Support Group (Intervention Group) | Control Group
Number analyzed (Participants) | 30 | 30
points
  Baseline | 36 (23.4) | 30.1 (19.2)
  Postintervention (6 months): number analyzed (Participants) | 29 | 30
  Postintervention (6 months) | 17.3 (12.5) | 34.3 (15.5)
  3 months follow-up (9 months): number analyzed (Participants) | 27 | 27
  3 months follow-up (9 months) | 16.5 (9.5) | 37 (15.8)

4. Secondary Outcome: Dementia Understanding of the Caregivers About Dementia
Description: The participant will be evaluated by the questionnaire originating from Northern Ireland Life and Time Survey questionnaire which includes 7 items. The score will range from 0 to 7. A higher score indicates a better outcome.
Time Frame: Baseline, post-intervention (6 months) and three-months follow-up (9 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Informational Support Group | Control Group
Number analyzed (Participants) | 30 | 30
points
  Baseline | 3.8 (1.5) | 3.5 (1.2)
  Postintervention: number analyzed (Participants) | 29 | 30
  Postintervention | 5.8 (1.3) | 2.9 (0.9)
  3 months follow-up: number analyzed (Participants) | 27 | 27
  3 months follow-up | 6.2 (1.3) | 3.1 (0.9)

5. Secondary Outcome: Phase 2: Perceived Social Support of the Caregivers
Description: The participant will be evaluated by the Multidimensional perceived social support scale (MSPSS) which includes 12 items. Each item is scored from 1 (very strongly disagree) to 7 (very strongly agree), based on a 7-point Likert scale. The minimum score is 12 and the maximum score is 84. Higher scores indicate higher degrees of perceived social support
Time Frame: Baseline, post-intervention (6 months), and three-month follow-up (9 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Information Support Group: The participants in the intervention group will be added to a chat room in the Zalo app, created and managed by one investigator, which is named The Dementia Caregiver Support group. Weekly, the investigator will post one of the eight topics identified in Phase 1. Before posting the information, the investigator will ask the participants what topic they would like to read and discuss the week after by voting the answer. The posted information will be based on evidence-based resources and consulted by geriatricians, the neurologist, and the psychologist who specialize in dementia. Immediately after posting the topic, one investigator will call the participants to ensure the participants read and understand the post. The chat group monitor will also collect the questions or comments from the carers who are encouraged to share feelings or experiences with relevant questions. Then the investigator will post the answers after consulting with the experts.
Arm/Group | Information Support Group | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 9.1 (3.7) | 8.9 (3.1)
  Postintervention: number analyzed (Participants) | 29 | 30
  Postintervention | 6.3 (2.9) | 9.8 (2.4)
  Three-month follow-up: number analyzed (Participants) | 27 | 27
  Three-month follow-up | 6.2 (2.4) | 9.7 (2.0)

6. Secondary Outcome: Phase 2: Perceived Burden
Description: The participants will be evaluated by the Zarit 4-item burden interview, including 4 items. Each item is scored from 1 to 4. The total score ranges from 0 to 16. A Higher score indicates a higher feeling of burden.
Time Frame: Baseline, post-intervention (6 months), and three-month follow-up (9 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Informational Support Group | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 9.1 (3.7) | 8.9 (3.1)
  Postintervention: number analyzed (Participants) | 29 | 30
  Postintervention | 6.2 (2.9) | 9.8 (2.4)
  Three-month follow-up: number analyzed (Participants) | 27 | 27
  Three-month follow-up | 6.2 (2.4) | 9.7 (2.0)

ADVERSE EVENTS:
Time Frame: 10 months
Description: In Phase 1, participants participated solely in qualitative interviews to describe their experiences and did not receive any intervention. As no intervention or experimental procedures were administered, there was no potential for harm or adverse events in this phase.
Groups:
- Phase 1: Qualitative Interviews: In-depth interviews were conducted to explore caregivers' knowledge and skill needs in providing care for people with dementia
Arm/Group | Phase 1: Qualitative Interviews | Phase 2: Informational Support Group (Intervention Group) | Phase 2: Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/20 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT04958707/Prot_SAP_000.pdf